CLINICAL TRIAL: NCT04287803
Title: Prehospital Analgesia in Adults Using Inhaled (PAIN) Methoxyflurane : A Feasibility Study
Brief Title: Prehospital Analgesia in Adults Using Inhaled Methoxyflurane : A Feasibility Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20191107100
Record Dates: First submitted 2019-12-02; First posted 2020-02-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pain, Acute; Trauma
Keywords: prehospital; paramedic; ambulance; methoxyflurane; Penthrox; Penthrane
MeSH Terms: conditions — Acute Pain; Wounds and Injuries | interventions — Methoxyflurane

STUDY DESIGN:
Intervention Model Description: Feasibility study to inform the multicentred prehospital prospective observational step wedge design trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention Arm (Experimental): Methoxyflurane will be introduced and data will be captured to inform future multicentred step wedge design study. (This study is a feasibility study)
  Interventions: Drug: Methoxyflurane

INTERVENTIONS:
Drug: Methoxyflurane — Methoxyflurane 3mls will be self administered by patients meeting the inclusion criteria with acute traumatic pain scores >=4
  Other Names: Penthrox; Penthrane

SUMMARY:
Pain is common and can contribute to both psychological and physiological effects if not treated. Currently primary care paramedics have limited selections within their pain management tool box. This contributes to inadequate pain management. Methoxyflurane is a safe, easy and effective choice in prehospital management of pain. The impact of this feasibility trial, will hope to inform the larger multi-centred trial and then support the implementation of out-of-hospital Canadian National Guidelines for prehospital pain control, enabling paramedics to provide rapid, effective prehospital pain relief to patients.

DETAILED DESCRIPTION:
This will be a single-centred prehospital prospective observational feasibility study to evaluate the ability to perform a multicentred step wedge design trial. The feasibility outcomes will provide evidence for the development of the multicentred study and will capture clinical metrics to inform this larger study. A waver of consent will be sought from the ethics board with participation consent for paramedics understanding the risk of using a gas for analgesia. Patient >= 18 years of age with traumatic pain with a verbal score >= to 4 will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* Acute pain from traumatic injury
* numeric pain score >=4

Exclusion Criteria:

* Allergy or sensitivity to methoxyflurane
* History or family history of malignant hyperthermia
* Pregnant or breast-feeding patients
* Known renal impairment
* Known liver disease
* Methoxyflurane use within previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Time to ethics approval for single site | from ethics submission up to 90 days
  Target: ,<= 3 months (90 days) from ethics submission
Time to readiness to initiate the clinical trial | From ethics approval up to 90 days
  Target, <= 3 months (90 days) from ethics approval
Evaluation of outcome data collected | For length of study, up to 100 patients
  Target: 100% of data captured in >90% cases
Study protocol compliance by paramedics | For length of study, up to 100 patients
  Target, >= 80%

SECONDARY OUTCOMES:
Verbal numeric pain rating score (0-10) initial and recorded every 5 minutes | For length of study, up to 100 patients specifically from patient contact to transfer of care in the emergency department
  Degree of change
Need for rescue medication (as defined by addition of any other pain medication after methoxyflurane administration, during paramedic care) | For length of study, up to 100 patients. specifically from patient contact to transfer of care in the emergency department
  If other medication are used to control pain
Transport time | For length of study, up to 100 patients, specifically departure scene to arrival at hospital
  Defined by departure from scene to arrival at hospital
Time to first administration of methoxyflurane | For length of study, up to 100 patients. Specifically time from patient contact to first inhalation of methoxyflurane
  Time from first patient contact to first inhalation of methoxyflurane
Vital signs and level of consciousness | From patient contact to transfer of care
  Vital signs including (Heart rate, Blood pressure, Respiratory rate, Oxygen saturation, Temperature, Glasgow Coma Scale (GCS))
Adverse events post administration of methoxyflurane: | For length of study, up to 100 patients. Specifically from patient contact to transfer of care
  Example: any advanced airway interventions, oxygen requirement (oxygen saturations <94%), drop in blood pressure by 40% and/or <90 systolic, complaints of nausea or vomiting, malignant hyperthermia reaction).

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Austin, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Dr Michael A Austin, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified data for primary and secondary outcome maybe available to share.